CLINICAL TRIAL: NCT05853497
Title: A Multi-Component Weight Loss Intervention to Improve Outcomes of Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: South Dakota State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00149595
Record Dates: First submitted 2023-03-06; First posted 2023-05-10 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Arthropathy of Knee; Obesity
Keywords: Total Knee Arthroplasty; Total Knee Replacement
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Control (No Intervention): Standard care
- Intervention (Experimental): Multi-component weight loss intervention
  Interventions: Behavioral: Multi-Component Weight Loss Intervention

INTERVENTIONS:
Behavioral: Multi-Component Weight Loss Intervention — The intervention group will receive weekly 1-on-1 health coaching with a very-low calorie nutrition plan prior to total knee replacement and a conventional weight maintenance nutrition plan after surgery.
  Arms: Intervention

SUMMARY:
Obesity, specifically BMIs ≥35 or 40 kg/m2, are associated with an increased probability of poor outcomes of Total Knee Arthroplasty (TKA) including increased pain, risk for infection, poor joint function, and increased rates of hospital readmissions. Several orthopedic and public health organizations recommend weight loss prior to TJA for individuals with overweight/obesity. However, empirical evidence suggesting the effectiveness of pre-surgical weight loss on surgical and functional outcomes of TKA is extremely limited and is based primarily on non-randomized observational studies. Thus, to gain further insight regarding the feasibility and potential effectiveness of pre-surgical weight loss on outcomes of TKA, the proposed pilot trial will randomize 30 patients (age 50-75 yrs., BMI 35<40 kg/m2) scheduled for TKA through The University of Kansas Health System Department of Orthopedics and Sports Medicine (KUOrtho) to a multi-component weight loss (3-mo. pre-TKA, very low-calorie diet) and maintenance intervention (3-mo. post TKA, conventional maintenance diet) or standard care control which will include no dietary or weight loss advice. The weight loss/maintenance interventions will include reduced energy intake or energy intake prescribed for weight loss maintenance, increased physical activity, and individual behavior counseling. Outcomes will be assessed 1) baseline, i.e., 3 mos. prior to surgery, 2) 3 mos. i.e., at the completion of the weight loss intervention prior to TKA, 3) within a minimum of 2 weeks post TKA, and 4) 3 mos. post-TKA, i.e., after completion of the weight maintenance intervention to assess the feasibility and effectiveness of a remotely delivered multi-component pre-TKA weight loss and a post-TKA weight maintenance intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age: 50-75 years
* BMI: 35 to ≤40 kg/m2
* Patient of KU Health System Department of Orthopedics and Sports Medicine (KUOrtho)meeting all requirements for TKA surgery.
* TKA surgical date scheduled ≥3 mos. from consent
* Own a Bluetooth enabled computer, tablet, or smart phone with the ability to join remote telehealth sessions and sync study self-monitoring devices.

Exclusion Criteria:

* Weight loss ≥10 pounds in previous 6 months
* Dairy/milk protein allergy
* Currently pregnant/breastfeeding or planning to become pregnant during the study
* Currently being treated for an eating disorder or history of an eating disorder diagnosis
* Pacemaker
* Current Cancer
* Diabetes Type 1 (insulin dependent)
* Hyperuricemia (untreated)
* Inflammatory bowel disease (active)
* Liver disease requiring protein restriction
* Myocardial infarction within last 3 months
* Abnormal ECG
* Renal insufficiency.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Participant Retention Feasibility | 6 Months
  Feasibility will be based on retention of ≥ 80% participants (i.e., <20% participant dropout).
Participant Attendance Feasibility | 6 Months
  Feasibility will be based on ≥ 80% attendance at behavioral counseling sessions.

SECONDARY OUTCOMES:
Knee and Lower Extremity Physical Function (OARSI Test) | 6 Months
  Knee and lower extremity function will be compared between study arms using the Osteoarthritis Research Society International (OARSI) physical function test battery.
Fat Mass (kg) | 6 Months
  Changes in fat mass (kg) will be compared between study arms using dual x-ray absorptiometry (DEXA)
Fat Free Mass (kg) | 6 Months
  Changes in fat free mass (kg) will be compared between study arms using dual x-ray absorptiometry (DEXA)
Body Weight (kg) | 6 Months
  Changes in body weight (kg) will be compared between study arms using a calibrated body weight scale.
Self reported knee function | 6 Months
  Self-reported knee function will be compared between study arms using the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire. Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Herrmann, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No